CLINICAL TRIAL: NCT00956657
Title: Improving Cardiac Rehabilitation Session Attendance Using the Self-Regulatory Model and Motivational Interviewing: A Randomised Controlled Trial
Brief Title: Improving Cardiac Rehabilitation Session Attendance: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Gavin Taylor, Clinical Psychologist, NHS Greater Glasgow & Clyde
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: 08/S0710/65
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2009-08

CONDITIONS: Cardiac Rehabilitation
Keywords: Randomised Controlled Trial; Adherence; Patient Participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Psychological Intervention Session — One-off session aimed at changing participants beliefs around illness control and consequences, applied using a motivational interviewing style.

SUMMARY:
Cardiac rehabilitation (CR) programmes typically offer patients with heart disease a long-term programme of medical evaluation, exercise, education and counseling. National guidelines have recognized the positive impact that attendance at CR can have following heart attacks, angina and other heart problems. Patients who attend such a programme have been shown to have reduced health problems. Despite this, research suggests that the use of these services is poor and that the majority of patients eligible for these programmes do not continue to attend after their first class. A range of factors have been associated with non-adherence to CR, including psychological factors such as people's beliefs about their illness. For example, patients with high levels of perceived control over their illness after a heart attack appear to be more likely to attend CR classes than those with low levels of perceived control. Such findings suggest that changing patients' illness beliefs, specifically those associated with illness control and illness consequences, could help to increase adherence to CR programmes. Increased adherence to CR could improve health outcomes for patients with cardiac illnesses. The present study is therefore investigating the effectiveness of a one-session psychological intervention, based on a theory called the Self-Regulatory Model, in altering beliefs about illness among patients starting cardiac rehabilitation. Participants will be randomly assigned to a treatment or a non-treatment group. It is hoped that those who receive the treatment session will attend more CR classes.

ELIGIBILITY:
Inclusion Criteria:

* Attending first cardiac rehabilitation class at one of three hospital sites
* Participants had to be over 18

Exclusion Criteria:

* Unable to read and understand English information sheet and consent form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin H Taylor, MA (Hons), Principal Investigator — NHS Greater Glasgow & Clyde
Locations (3):
- United Kingdom (3):
  - Southern General Hospital, Glasgow
  - Stobhill Infirmary, Glasgow
  - Victoria Infirmary, Glasgow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in November 2008 and was completed in May 2009. All recruitment took place in out-patient cardiac rehabilitation departments within hospital buildings.
Groups:
- Treatment Group: Single treatment session provided by study PI. Session aimed to change participant illness beliefs using motivational interviewing techniques in order to improve adherence to cardiac rehabilitation classes.
- Treatment As Usual: Control group. Treatment received as usual.
Period: Overall Study
Arm/Group | Treatment Group | Treatment As Usual
Started | 18 | 13
Completed | 18 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Treatment As Usual | Total
Number analyzed (Participants) | 18 | 13 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 6 | 4 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (9.6) | 61 (10.6) | 62 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18 | 13 | 31

OUTCOME MEASURES:

1. Secondary Outcome: Illness Perceptions Questionnaire-Revised Scores
Description: Eight sub-scale scores obtained. Sub-scales include; Illness consequences, Illness Control, Treatment Control, Illness Identity, Emotional Representation, Illness Cause, Illness Coherence, Timeline Cyclical. Minimum and Maximum scores vary for each sub-scale.
Time Frame: 3-months after consent
Reporting Status: Not Posted
Measure: Number; unit: Units on a scale

2. Primary Outcome: CR Adherence
Description: Number of cardiac rehabilitation classes attended in total.
Time Frame: Approximately 3-months after recruitment
Measure: Mean (Standard Deviation); unit: Classes Attended
Arm/Group | Treatment Group | Treatment As Usual
Number analyzed (Participants) | 18 | 13
Classes Attended | 16.0 (5.2) | 14.4 (6.2)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/13
Other Adverse Events (participants affected / at risk) | 0/18 | 0/13

LIMITATIONS AND CAVEATS:
The small sample size of this study does not allow definitive conclusions to be drawn about the success or failure or this intervention approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No